CLINICAL TRIAL: NCT00384683
Title: Endothelial Dysfunction As A Predictor Of Perioperative Outcome In Major Thoracic Surgery - An Observational Study
Brief Title: Endothelial Dysfunction As A Predictor Of Perioperative Outcome
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-0434
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Endothelial Dysfunction
Keywords: Endothelial Dysfunction; Endothelial Cells; Perioperative Outcome; Blood Sample

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected to measure number of circulating blood cells that become endothelial cells. During surgery a small sample of lung tissue collected, if available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endothelial Dysfunction: Participants are scheduled for major chest (lung or esophagus) surgery or are a healthy volunteer. A blood test will quantify the number of cells that are destined to become endothelial cells.

SUMMARY:
The goal of this clinical research study is to learn whether the inability of certain blood vessel cells (endothelial cells) to function properly may help researchers to predict who is at risk for complications after surgery and whether this dysfunction contributes to complications after surgery. This study will use a blood test to quantify the number of cells that are destined to become endothelial cells.

DETAILED DESCRIPTION:
A small group of patients (about 12 out of every 100) are at risk of developing complications, for example lung infection, after their surgery. Researchers do not always know which patient is at risk or the reason why some patients develop these complications. Your participation in this study may help researchers to understand who is at risk and also the mechanism of some of the complications.

The inner layer of cells of blood vessels are called endothelial cells. This layer of cells plays a vital role in the normal function of blood vessels, including blood clotting and inflammation. Certain conditions, such as aging, smoking, high cholesterol, and some chemotherapies cause these cells to not function properly. Researchers can test whether these cells function properly by doing two simple tests - one is a blood test and the other uses ultrasound and temperature probes on the finger to look at the ability of arm blood vessels to dilate (expand).

The way your cells function will be tested within a month before your scheduled chemotherapy / radiation (if applicable), and again within a month before your major chest surgery. This will be done on those patients with surgery planned or scheduled.

About 2 tablespoons of blood will be drawn to measure the number of circulating blood cells that become endothelial cells.

During your scheduled surgery, the researcher will also collect just over a teaspoon of blood at the beginning of the surgery for an additional endothelial risk assessment and a small sample of lung tissue, if available. Tissue removed during long surgery is usually thrown away if it is not needed for diagnosis and or treatment purposes. The lung tissue sample collected for this research study will only be taken from lung tissue that is to be discarded. The lung tissue will be used to determine the amount of a naturally occurring substance thought to play a role in recruiting blood cells to repair injured lung tissue.

Blood samples (about 2 tablespoons) will also be collected after exercise, during your surgery, 24 hours after your surgery, and at 5 days after surgery or the time you discharge from the hospital (which ever is shorter). These blood samples will also be collected at your routinely schedule post operative clinic visits at 1 month, 6 months, and 1 year after surgery. The samples will be used to determine the amount of endothelial cells in the blood stream.

For healthy volunteers, blood samples (about 2 tablespoons) will be collected at baseline (prior to exercising), 15-30 minutes past peak exercise, 3 hours past peak exercise and at 24 hours past past peak exercise.

Data will be collected on you for 30 days after your surgery, and during the 1 year follow-up. These data will then be matched with the amount of cell function as measured before surgery to see if these tests may be used to help predict which patients are at increased risk for complications. No other measurements will be done and this study will not change your surgical procedure or lengthen your hospital stay.

This is an investigational study. About 90 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center (MDACC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for major thoracic surgery (lobectomy, pneumonectomy, esophagectomy).
2. Patients 18 years of age or older.
3. Patients who have signed the consent form to participate in the study.
4. Patients must have been evaluated in the Preanesthesia Clinic or by a staff Anesthesiologist preoperatively.
5. All laboratory and diagnostic evaluations required or used to evaluate the patient in the Preanesthesia Clinic must be completed. All patients must be approved for surgery by the standards of the Preanesthesia Clinic.

Exclusion Criteria:

1. Refusal to participate in the study.
2. Patient is under age 18.
3. Patient is unwilling to sign consent.
4. Patient is unable to exercise (bedridden or wheel chair bound).
5. Patient is enrolled in another study deemed by the investigator to affect oxygen metabolic efficiency and not presently the standard of care at MDACC.
6. Any patient whose condition is deemed unsatisfactory for surgery after the preanesthetic evaluation.
7. Surgery canceled for any reason. The patient may reenter the study if surgery is rescheduled.
8. Patient has had a myocardial infarction within 3 months of visiting the Preanesthesia Clinic or presents with new or unstable angina.
9. Patient has a history of cerebrovascular accident or transient ischemic attacks within 3 months of visiting the Preanesthesia Clinic.
10. Patient has a history of pulmonary embolic event within 3 months of visiting the Preanesthesia Clinic.
11. Patient known to have acute or chronic deep vein thrombosis.
12. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants is scheduled to have major chest (lung or esophagus) surgery or is a healthy volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Number of Patient Major Pulmonary Events (MPE) | Baseline (entry in study) to end of study (estimated 1 year post-operative)

SECONDARY OUTCOMES:
Patient's Duration of intensive care unit / hospital length of stay | Baseline to final day of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Reza-John Mehran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Official Web Site — http://www.mdanderson.org